CLINICAL TRIAL: NCT02664935
Title: National Lung Matrix Trial: Multi-drug, Genetic Marker-directed, Non-comparative, Multi-centre, Multi-arm Phase II Trial in Non-small Cell Lung Cancer
Brief Title: National Lung Matrix Trial: Multi-drug Phase II Trial in Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Cancer Research UK (Other); AstraZeneca (Industry); Pfizer (Industry); Experimental Cancer Medicine Centres (Other); Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_14-072; 2014-000814-73 (EudraCT Number); ISRCTN38344105 (Other: ISRCTN Registry)
Record Dates: First submitted 2016-01-05; First posted 2016-01-27 (Estimated); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer; Carcinoma, Squamous Cell; Adenocarcinoma
Keywords: NSCLC; Lung Cancer; Adenocarcinoma; Matrix; SMP2; Umbrella Trial Design; Multi-arm
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell; Adenocarcinoma; Lung Neoplasms | interventions — AZD4547; vistusertib; palbociclib; Crizotinib; AZD 6244; Docetaxel; capivasertib; osimertinib; durvalumab; sitravatinib; ceralasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Arm A: AZD4547 (Experimental): AZD4547 - FGFR Inhibitor Route & Formulation: Oral, Tablets Strengths: 20 & 80mg Trial Dose & Schedule: 80 mg BD, Continuous dosing, 21 day cycle.
  Interventions: Drug: AZD4547
- Arm B: Vistusertib (AZD2014) (Experimental): Vistusertib (AZD2014) - MTORC1/2 Inhibitor Route & Formulation: Oral, Tablets Strengths: 25mg Trial Dose & Schedule: 125 mg BD, Intermittent dosing (2 continuous days in 7), 28 day cycle.
  Interventions: Drug: Vistusertib
- Arm C: Palbociclib (Experimental): Palbociclib - CDK4/6 Inhibitor Route & Formulation: Oral, Capsules Strengths: 75, 100 & 125mg Trial Dose & Schedule: 125 mg OD, Intermittent dosing (21 days on, 7 days off), 28 day cycle.
  Interventions: Drug: Palbociclib
- Arm D: Crizotinib (Experimental): Crizotinib - ALK Inhibitor Route & Formulation: Oral, Capsules Strengths: 200 & 250mg Trial Dose & Schedule: 250 mg BD, Continuous dosing, 21 day cycle.
  Interventions: Drug: Crizotinib
- Arm E: Selumetinib & Docetaxel (Experimental): AZD6244 (Selumetinib) - MEK Inhibitor Route & Formulation: Oral, Capsules Strengths: 25mg Trial Dose & Schedule: 75 mg BD, Continuous dosing, 21 day cycle.
  Docetaxel - Chemotherapy Route & Formulation: IV infusion over 30-60 minutes, concentrate for solution for infusion.
  Trial Dose & Schedule: 75 mg/m2, 3-weekly, 21 day cycle.
  Interventions: Drug: Selumetinib; Drug: Docetaxel
- Arm F: AZD5363 (Experimental): AZD5363 - AKT Inhibitor Route & Formulation: Oral, Tablets Strengths: 80 & 200mg Trial Dose & Schedule: 480 mg BD, Intermittent dosing (4 days on, 3 days off), 28 day cycles.
  Interventions: Drug: AZD5363
- Arm G: Osimertinib (AZD9291) (Experimental): Osimertinib (AZD9291) - EGFRM+ and T790M+ Inhibitor Route & Formulation: Oral, Tablets Strengths: 80mg Trial Dose & Schedule: 80 mg OD, Continuous dosing, 21 day cycles.
  Interventions: Drug: Osimertinib
- Arm NA: Durvalumab (MEDI4736) (Experimental): Durvalumab (MEDI4736) - Anti-PDL1 Route & Formulation: IV Infusion, Lyophilized powder for solution for infusion Strengths: Vial containing 200mg Trial Dose & Schedule: 10 mg/kg IV, 2-weekly.
  Interventions: Drug: Durvalumab
- Arm H: Sitravatinib (Experimental): Sitravatinib - VEGFR Inhibitor Route & Formulation: Oral, Capsules Strengths: 10 & 40mg Trial Dose & Schedule: 120 mg OD, Continuous dosing, 21 day cycles.
  Interventions: Drug: Sitravatinib
- Arm J: AZ6738 & Durvalumab (Experimental): AZD6738 - ATR Inhibitor Route & Formulation: Oral, Tablets Strengths: 20mg, 80mg, 100mg Trial Dose & Schedule: 240 mg twice daily (BD) on days 15-28 of 28 day cycle.
  Durvalumab (MEDI4736) - Anti-PDL1 Route & Formulation: IV Infusion, Lyophilized powder for solution for infusion Strengths: Vial containing 500mg Trial Dose & Schedule: 1500mg on day 1 of each 28 day cycle
  Interventions: Drug: Durvalumab; Drug: AZD6738

INTERVENTIONS:
Drug: AZD4547 — FGFR Inhibitor
  Arms: Arm A: AZD4547
Drug: Vistusertib — MTORC1/2 Inhibitor
  Other Names: AZD2014
  Arms: Arm B: Vistusertib (AZD2014)
Drug: Palbociclib — CDK4/6 Inhibitor
  Arms: Arm C: Palbociclib
Drug: Crizotinib — ALK/MET/ROS1 Inhibitor
  Arms: Arm D: Crizotinib
Drug: Selumetinib — MEK Inhibitor
  Other Names: AZD6244
  Arms: Arm E: Selumetinib & Docetaxel
Drug: Docetaxel — Taxane, anti-mitotic cytotoxic chemotherapy
  Arms: Arm E: Selumetinib & Docetaxel
Drug: AZD5363 — AKT Inhibitor
  Arms: Arm F: AZD5363
Drug: Osimertinib — EGFRm+ T790M+ Inhibitor
  Other Names: AZD9291
  Arms: Arm G: Osimertinib (AZD9291)
Drug: Durvalumab — Anti-PDL1
  Other Names: MEDI4736
  Arms: Arm J: AZ6738 & Durvalumab; Arm NA: Durvalumab (MEDI4736)
Drug: Sitravatinib — VEGFR Inhibitor
  Other Names: MGCD516
  Arms: Arm H: Sitravatinib
Drug: AZD6738 — ATR inhibitor
  Arms: Arm J: AZ6738 & Durvalumab

SUMMARY:
The trial consists of a series of parallel multi-centre single arm phase II trial arms, each testing an experimental targeted drug in a population stratified by multiple pre-specified actionable target putative biomarkers. The primary objective is to evaluate whether there is a signal of activity in each drug-(putative)biomarker cohort separately. A Bayesian adaptive design is adopted to achieve this objective and statistical details are given in the Protocol.

DETAILED DESCRIPTION:
The trial is primarily an enrichment putative biomarker design, including patients who are positive for at least one of the actionable targets included in the trial. Patients who are positive for just one putative biomarker will receive the experimental targeted drug specific for that putative biomarker. Putative biomarkers within each drug cohort have been chosen such that in the majority of cases it is not expected that patients will be positive for two or more putative biomarkers within the same drug. In the rare situation that patients are positive for two or more putative biomarkers relevant across different drugs, treatment will be allocated in accordance with the following strategy:

* All amplifications and rearrangements will be treated with targeted agent appropriate to them irrespective of concomitant mutations. This will yield crucial predictive biomarker information.
* For concomitant mutations decisions will be made by the Chief Investigator on a case-by-case basis and based on close consideration of pathway preference and likely dominance of one signal pathway over another together with any pre-clinical efficacy studies that address the activity of the drugs in the presence of concomitant mutations. A trumping strategy has been devised for this purpose.

ELIGIBILITY:
Core inclusion and exclusion criteria are presented below. Additional inclusion/exclusion criteria apply to each arm and are presented in the relevant arm supplements of the protocol.

Inclusion Criteria:

* Prior anti-cancer treatment:

  * Patients who refuse any standard of care first line therapy, are eligible to receive National Lung Matrix Trial treatment as first line therapy, providing they explicitly consent to this effect.
  * Patients who have previously consented to and received standard of care first line therapy must have completed all standard of care therapy that the treating oncologist thinks is appropriate. As a minimum patients must have failed one or more lines of treatment (either radiological documentation of disease progression or due to toxicity). Patients whose disease has increased in size but is not classed as progressive disease as per RECIST criteria, will be eligible. Patients with no change at all in dimension of disease (i.e. true stability) after first line therapy will not be eligible.
  * Patients who have progressed after surgical resection and adjuvant therapy will be eligible for entry without the need for the administration of first line metastatic therapy.
  * Patients will also be eligible without the necessity for first line regimen if they have relapsed within 6 months of completion of definitive chemoradiation.
* Consented and provided an adequate specimen to adequately characterise the molecular genotype of the tumour in the molecular pre-screening according to the molecular exclusion rules (see Section 6.4 for definition of an adequate sample).
* Histological or cytologically confirmed NSCLC stage III (not suitable for radical radiotherapy or surgery) or stage IV. This includes patients who may have abnormal histology, but IHC strongly support either squamous cell carcinoma (p63 positivity) or adenocarcinoma (Thyroid transcription factor 1 [TTF1] positivity). If a physician and pathologist are convinced after multi-disciplinary review that the patient has stage III or IV NSCLC but where all the IHC is negative and the morphology does not distinguish a specific sub-type, these patients will be eligible for non-histology specific cohorts.
* CT or MRI scan of head, chest and abdomen within 28 days of treatment demonstrating measurable disease as per RECIST version 1.1 (see Appendix 1: Response Evaluation Criteria in Solid Tumours Version 1.1). (The same imaging modality must be used throughout treatment).
* Adequate haematological function within 7 days of treatment.

  * Haemoglobin ≥ 90 g/L.
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
  * Platelets ≥ 100 x 109/L.
* Adequate hepatic function within 7 days of treatment in patients with no liver metastasis (see arm specific entry criteria for adequate hepatic function in patients with liver metastases).

  * Total serum bilirubin ≤ 1.5 x upper limit of normal (ULN). (Note that this will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of evidence of haemolysis or hepatic pathology), who may be allowed inclusion at the discretion of the local Investigator).
  * Alanine transferase (ALT) ≤ 2.5 x ULN.
  * Aspartate transferase (AST) ≤ 2.5 x ULN.
* Adequate renal function within 7 days of treatment.

  * Creatinine clearance (CLcr) >50 ml/min (measured or calculated by Cockcroft and Gault equation - see Appendix 4: Cockcroft Gault Formula - Creatinine Clearance). If calculated CLcr is <50 ml/min a direct measurement of glomerular filtration rate (GFR) such as EDTA may be performed. If the value is >50 ml/min the patient is eligible.
* Age ≥ 18 years.
* Females must agree to use adequate contraceptive measures (as defined in Section 6.3), should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

  * Post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
  * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
  * Women aged under 50 years old would be consider postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range for the institution.
* Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses.

Exclusion Criteria:

* Major surgery (excluding placement of vascular access) within 4 weeks prior to treatment.
* Nausea, vomiting, chronic gastrointestinal diseases (e.g. inflammatory bowel disease) that would preclude adequate absorption.
* Any psychological, familial, sociological or geographical condition hampering protocol compliance.
* Concurrent malignancies or invasive cancers diagnosed within past 3 years except for adequately treated basal cell carcinoma of the skin and in situ carcinoma of the uterine cervix.
* Judgement by the local Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
* Any unresolved toxicity of grade 2, 3 or 4 from previous treatment (excluding alopecia) at Registration (see CTCAE - Appendix 3: Common Toxicity Criteria Gradings).
* Patients who have previous symptomatic brain metastases or spinal cord compression are excluded unless they have had adequate treatment, no evidence of progression or symptoms, and have had no requirement for steroid treatment in the previous 28 days before commencement of trial treatment.
* Patients with asymptomatic brain metastases picked up at screening CT scan are not excluded providing that in the view of the local Investigator they do not require immediate radiotherapy or surgical intervention, and have had no requirement for steroid treatment in the previous 28 days before commencement of trial treatment.
* As judged by the local Investigator, any evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus. Screening for chronic conditions is not required.
* Pregnant and lactating patients (patients of childbearing potential must have a negative pregnancy test prior to registration).

Cardiac exclusion criteria, performance status and prior treatment washout periods are detailed within the National Lung Matrix Trial arm-specific eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Objective response (OR) | From baseline until disease progression, assessed up to 18 months.
  CT scans every 6 weeks from baseline until disease progression (Primary outcome for all Trial Arms except Arm C). Investigators expect patients to participate in the study for a maximum of 18 months, however cannot guarantee that some patients may participate over 18 months.
Progression-free survival time (PFS) | From date of commencement of trial treatment to date of CT scan when progressive disease first recorded or date of death without previously recorded progression, assessed up to 18 months.
  Defined as the time from commencement of trial treatment to the date of CT scan when progressive disease first recorded or date of death without previously recorded progression (Primary Outcome for Arm C only). Patients who are alive with no recorded progression at the time of analysis will be censored at the date of the CT scan when they were last recorded with an evaluable measure that was not progression. Investigators expect patients to participate in the study for a maximum of 18 months, however, cannot guarantee that some patients may participate over 18 months.
Durable clinical benefit (DCB) | From baseline until the first scan after 24 weeks showing the patient free of disease progression.
  A patient will be defined as experiencing DCB if they remain free of disease progression at their fourth CT or MRI scan since treatment start date, i.e. approximately 24 weeks, or at any scan after 24 weeks that shows the patient free of disease progression (co-primary outcome for all Trial Arms except Arm C & G)

SECONDARY OUTCOMES:
Best percentage change in sum of target lesion diameters (PCSD) | From baseline until disease progression, assessed up to 18 months.
  At each evaluation, the longest diameters of all selected target lesions will be measured and summed and the percentage change from the baseline measurement will be calculated. The best percentage change is the one that reflects either the greatest decrease or the least increase over the whole period of assessment. Investigators expect patients to participate in the study for a maximum of 18 months, however cannot guarantee that some patients may participate over 18 months.
Time to Progression (TTP) | The time from commencement of trial treatment to the date of the CT scan when progressive disease first recorded, assessed up to 18 months.
  This is defined as the time from commencement of trial treatment to the date of the CT scan when progressive disease first recorded. Patients with no recorded progression at the time of analysis or who die without recorded progression will be censored at the date of the CT scan when they were last recorded with an evaluable measure that was not progression. Investigators expect patients to participate in the study for a maximum of 18 months, however cannot guarantee that some patients may participate over 18 months.
Overall survival time (OS) | From time of commencement of trial treatment until date of death, assessed up to 18 months.
  This is defined as the time of commencement of trial treatment to the date of death. Patients who are alive at the time of analysis will be censored at the date last seen alive. Investigators expect patients to participate in the study for a maximum of 18 months, however cannot guarantee that some patients may participate over 18 months.
Adverse Events (AE) | From date of informed consent to trial treatment until 28 days after the last administration of the last treatment, assessed up to 18 months.
  Adverse events will be recorded in relation to each cycle of treatment and graded according to Common Terminology Criteria for Adverse Events (CTCAE). The incidence of each adverse event (all grades and grade 3/4) will be reported as a per-patient-cycle rate and as a per-patient rate. Investigators expect patients to participate in the study for a maximum of 18 months, however cannot guarantee that some patients may participate over 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Gary W Middleton, Principal Investigator — University of Birmingham
Locations (25):
- United Kingdom (25):
  - Aberdeen Royal Infirmary, Aberdeen
  - Belfast City Hospital, Belfast Health and Social Care Trust, Belfast
  - Queen Elizabeth Hospital Birmingham, University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Birmingham Heartlands Hospital, Heart of England NHS Foundation Trust, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Addenbrooke's Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Velindre Cancer Centre, Velindre NHS Trust, Cardiff
  - Colchester General Hospital, Colchester
  - Edinburgh Cancer Centre, Western General Hospital, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St. James' University Hospital, Leeds Teaching Hospital NHS Trust, Leeds
  - Leicester Royal Infirmary, University Hospitals of Leicester NHS Trust, Leicester
  - Royal Marsden Hospital, The Royal Marsden NHS Foundation Trust, London
  - Charing Cross Hospital, Imperial College Healthcare NHS Trust, London
  - Guy's Hospital, Guy's and St Thomas' NHS Foundation Trust, London
  - St Bartholomew's Hospital, Barts Health NHS Trust, London
  - University College Hospital, University College London Hospitals NHS Foundation Trust, London
  - Maidstone Hospital, Maidstone
  - The Christie Hospital, The Christie NHS Foundation Trust, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Sir Bobby Robson Cancer Trial Research Centre, The Newcastle upon Tyne Hospitals, Newcastle
  - Churchill Hospital, Oxford University Hospitals NHS Foundation Trust, Oxford
  - Weston Park Hospital, Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Southampton General Hospital, University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Middleton G, Crack LR, Popat S, Swanton C, Hollingsworth SJ, Buller R, Walker I, Carr TH, Wherton D, Billingham LJ. The National Lung Matrix Trial: translating the biology of stratification in advanced non-small-cell lung cancer. Ann Oncol. 2015 Dec;26(12):2464-9. doi: 10.1093/annonc/mdv394. Epub 2015 Sep 25. PMID 26410619
- [Result] Middleton G, Fletcher P, Popat S, Savage J, Summers Y, Greystoke A, Gilligan D, Cave J, O'Rourke N, Brewster A, Toy E, Spicer J, Jain P, Dangoor A, Mackean M, Forster M, Farley A, Wherton D, Mehmi M, Sharpe R, Mills TC, Cerone MA, Yap TA, Watkins TBK, Lim E, Swanton C, Billingham L. The National Lung Matrix Trial of personalized therapy in lung cancer. Nature. 2020 Jul;583(7818):807-812. doi: 10.1038/s41586-020-2481-8. Epub 2020 Jul 15. PMID 32669708
- See also: PL02.09 National Lung Matrix Trial (NLMT): First Results from an Umbrella Phase II Trial in Advanced Non-Small Cell Lung Cancer (NSCLC) Middleton, G. et al. Journal of Thoracic Oncology, Volume 14, Issue 10, S7 — https://doi.org/10.1016/j.jtho.2019.08.060
- See also: MA06. 06 A Phase II Trial of Ceralasertib and Durvalumab in Advanced Non-Small Cell Lung Cancer (NSCLC) with and without RAS Mutations: Results of NLMT Arm J — https://doi.org/10.1016/j.jtho.2023.09.154
- Available data/document: Trial Website — https://www.birmingham.ac.uk/research/crctu/trials/lung-matrix/index.aspx